CLINICAL TRIAL: NCT00345878
Title: Phase 3, Open, Age-stratified Study to Assess Immunogenicity and Safety of GSK Biologicals' HPV-16/18 Vaccine Administered Intramuscularly According to 3-dose Schedule (0,1,6 Months) in Healthy Female Subjects Aged 15 - 55 Years and Long Term Follow-up
Brief Title: Study to Evaluate the Immune Response and Safety of GSK Biologicals' HPV Vaccine in Healthy Women Aged 18-35 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 105926
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Results first posted 2009-12-15 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2016-11

CONDITIONS: Infections, Papillomavirus
Keywords: HPV-16/18 L1 VLP AS04; Cervical neoplasia; Cervical cancer; Human Papillomavirus (HPV); Double-blind; AS04
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Cervarix Group (Experimental): Subjects received 3 doses of HPV-16/18 L1 VLP AS04 (Cervarix™) according to a 0, 1, 6-month schedule.
  Interventions: Biological: HPV-16/18 L1 VLP AS04 (Cervarix TM)
- Placebo Group (Placebo Comparator): Subjects received 3 doses of Placebo according to a 0, 1, 6-month schedule.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — Three doses of vaccine administered intramuscularly according to a 0, 1, 6-month schedule.
  Arms: Placebo Group
Biological: HPV-16/18 L1 VLP AS04 (Cervarix TM) — Three doses of vaccine administered intramuscularly according to a 0, 1, 6-month schedule.
  Other Names: GSK Biologicals' HPV-16/18 VLP/AS04 vaccine
  Arms: Cervarix Group

SUMMARY:
Human papillomavirus infection has clearly been recognized as the cause of cervical cancer. The infection of the cervix by certain oncogenic types of HPV, if not cleared, can lead to cervical cancer in women. This study will evaluate the immunogenicity and safety of the HPV-16/18 L1 VLP AS04 vaccine.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
The protocol was primarily amended for the following reasons:

* Merck's tetravalent HPV vaccine, Gardasil®, has been licensed and is now becoming commercially available in an increasing number of countries. Therefore, the study procedures were revised to include questions at every visit to determine if subjects have received an HPV vaccine outside of the study.
* It was decided to offer GSK Biologicals' HPV vaccine to all subjects in the control group at the end of the study. The HPV vaccine will be offered to these subjects based on its local indication once the vaccine is marketed in Malaysia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A female from Malaysia between, and including, 18 and 35 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects must have a negative urine pregnancy test.
* Subjects of childbearing potential at the time of study entry must be abstinent or must be using an effective method of birth control for 30 days prior to vaccination and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after the first dose of vaccine. Administration of routine vaccines up to 8 days before the first dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* previous administration of components of the investigational vaccine
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Hypersensitivity to latex.
* Acute disease at the time of enrolment.
* Known acute or chronic, clinically significant neurologic, pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* History of chronic condition(s) requiring treatment.
* Administration of immunoglobulins and/or any blood product within three months preceding the first dose of study vaccine(s) or planned administration during the study period. Enrolment will be deferred until the subject is outside of specified window.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2006-09-25; Primary Completion 2007-12-21 (Actual); Study Completion 2007-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Malaysia (2):
  - GSK Investigational Site, Kerajaan Persekutuan Putrajaya
  - GSK Investigational Site, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 105926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 105926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cervarix Group | Placebo Group
Started | 135 | 136
Completed | 131 | 135
Not Completed | 4 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Placebo Group | Total
Number analyzed (Participants) | 135 | 136 | 271
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.8 (3.91) | 25.0 (4.14) | 24.9 (4.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 136 | 271
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Seroconverted for Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies
Description: Seroconversion is defined as the appearance of antibodies with titers greater than or equal to the predefined cut-off value in the serum of subjects seronegative before vaccination. Cut-off values assessed include 8 enzyme-linked immunosorbent assay units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: At Month 7
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 112 | 115
Participants
  Anti-HPV16 | 112 | 4
  Anti-HPV18: number analyzed (Participants) | 106 | 113
  Anti-HPV18 | 106 | 2

2. Secondary Outcome: Titers of Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as Enzyme-linked Immunosorbent Assay Units Per Milliliter (EL.U/mL).
Time Frame: At Month 0 and Month 7
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 126 | 129
EL.U/mL
  Anti-HPV16 (at Month 0) | 5.1 [4.3 to 6.0] | 4.6 [4.2 to 5.0]
  Anti-HPV16 (at Month 7): number analyzed (Participants) | 126 | 127
  Anti-HPV16 (at Month 7) | 11133.3 [9817.6 to 12625.3] | 4.7 [4.2 to 5.3]
  Anti-HPV18 (at Month 0): number analyzed (Participants) | 122 | 127
  Anti-HPV18 (at Month 0) | 4.3 [3.9 to 4.7] | 4.2 [3.8 to 4.7]
  Anti-HPV18 (at Month 7): number analyzed (Participants) | 122 | 127
  Anti-HPV18 (at Month 7) | 4264.2 [3771.6 to 4821.2] | 4.2 [3.8 to 4.7]

3. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Solicited general symptoms assessed include arthralgia, fatigue, fever, gastro-intestinal symptoms, headache, myalgia, rash and urticaria.
Time Frame: During the 7 days after each vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 132 | 135
Participants
  Pain | 121 | 101
  Redness | 48 | 40
  Swelling | 42 | 25
  Arthralgia | 39 | 26
  Fatigue | 52 | 48
  Fever (above 37.5 degree Celsius) | 19 | 17
  Gastro-intestinal symptoms | 18 | 18
  Headache | 46 | 47
  Myalgia | 48 | 32
  Rash | 4 | 7
  Urticaria | 4 | 2

4. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited adverse event = Any adverse event (AE) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: Within 30 days after any vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 135 | 136
Participants | 30 | 36

5. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events as New Onset Chronic Diseases (NOCDs) and Other Medically Significant Adverse Events (AEs)
Description: NOCDs assessed include e.g. autoimmune disorders, asthma, type I diabetes, allergies,...
  Medically significant AEs assessed include AEs prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or SAEs that are not related to common diseases.
Time Frame: Throughout the study period (up to Month 7)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 135 | 136
Participants
  NOCDs | 1 | 0
  Medically significant AEs | 10 | 11

6. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: Serious adverse events assessed include medical occurrences that results in death, is life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Throughout the study period (up to Month 7)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 135 | 136
Participants | 3 | 3

ADVERSE EVENTS:
Description: Events collected by systematic assessment are reported for subjects with a symptom diary card available.
  Events collected by a non-systematic method are reported for the Total Vaccinated cohort.
Arm/Group | Cervarix Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 3/135 | 3/136
Other Adverse Events (participants affected / at risk) | 126/135 | 114/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=135) | Placebo Group (N=136)
Dengue fever (Infections and infestations) | 1 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Chronic tonsillitis (Infections and infestations) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=135) | Placebo Group (N=136)
Pain (General disorders) | 121 | 101
Redness (General disorders) | 48 | 40
Swelling (General disorders) | 42 | 25
Arthralgia (General disorders) | 39 | 26
Fatigue (General disorders) | 52 | 48
Fever (above 37.5 degree Celsius) (General disorders) | 19 | 17
Gastro-intestinal symptoms (General disorders) | 18 | 18
Headache (General disorders) | 46 | 47
Myalgia (General disorders) | 48 | 32
Rash (General disorders) | 4 | 7
Upper respiratory tract infection (Infections and infestations) | 8 | 10
Influenza (Infections and infestations) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.